CLINICAL TRIAL: NCT02115919
Title: Phase 1 Study of Multikine in the Treatment of Perianal Warts
Brief Title: Safety Study of Multikine in the Treatment of Perianal Warts
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll prospective subject for dose escalation
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: CEL-SCI Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2013.0080
Record Dates: First submitted 2013-08-15; First posted 2014-04-16 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Condyloma
Keywords: condyloma; HIV
MeSH Terms: conditions — Condylomata Acuminata | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): Cohort A participants will undergo perilesional Multikine injections (200IU) once daily, Monday through Friday, for 14 days, off for 14 days, then again once daily, Monday through Friday for 14 days.
  Interventions: Drug: Leukocyte Interleukin, Injection 200IU
- Cohort B (Experimental): Cohort B participants will undergo perilesional Multikine injections 400IU once daily, Monday through Friday, for 14 days, off for 14 days, then again once daily, Monday through Friday for 14 days.
  Interventions: Drug: Leukocyte Interleukin, injection 400IU

INTERVENTIONS:
Drug: Leukocyte Interleukin, Injection 200IU — Cohort A participants will receive 200IU Multikine perilesional injections once daily, Monday through Friday, for 14 days, then 14 days off with out any Multikine injections received. After the 14 days without receiving the Investigational Product injections they will begin a second round of 200IU Multikine perilesional injections once daily, Monday through Friday for 14 days.
  Other Names: Multikine, Injection 200IU
  Arms: Cohort A
Drug: Leukocyte Interleukin, injection 400IU — Cohort B participants will receive 400IU Multikine perilesional injections once daily, Monday through Friday, for 14 days, then they will not receive any Multikine perilesional injections for 14 days. After the 14 day rest period when the participants did not receive the Investigational Product injections they will begin a second round of 400IU Multikine perilesional injections every day, Monday through Friday, for 14 days.
  Other Names: Multikine, Injection 400IU
  Arms: Cohort B

SUMMARY:
Caused by the human papillomavirus (HPV), anogenital warts are a common sexually-transmitted infection (STI). They are distressing to those who have them and are a source of viral shedding and transmission to others. Treatment of warts is aimed at destruction of the lesion.

Objectives:

1. Establish safety of Multikine in treatment of perianal condyloma.
2. Describe presence of anal HPV and anal dysplasia in participants with perianal condyloma.
3. Describe adverse effects associated with Multikine in the management of perianal condyloma.

Design:

Phase I, dose-escalation trial. Potential participants desiring treatment for their perianal warts will be referred to study by their primary clinician. All participants will undergo baseline anal Pap, anal HPV subtyping, perianal condyloma characterization (count, measurement, photography), and complete a baseline questionnaire. Cohort A participants will undergo perilesional Multikine injections (200IU) once daily, Monday through Friday, for 14 days, off for 14 days, then again once daily, Monday through Friday for 14 days. If no serious adverse events are noted after 4 weeks of therapy, cohort B will be studied using the same schedule but with a dose of 400IU per treatment. Each participant will undergo anal Pap and anal HPV subtyping once weekly during treatment. Condyloma characterization (count, measurement, photography) will occur prior to each treatment. After treatment completed, participants will complete a follow-up visit at 70, 100, 130, 160 days and have anal Pap, anal HPV subtyping, and perianal condyloma characterization (count, measurement, photography) performed.

Subjects:

The study will be open to adult men and women who are HIV-infected who receive medical care from the Naval Medical Center San Diego.

Main Outcome Measures:

1. Perianal wart characterization [count, measurement (in millimeters diameter)], photography)
2. HPV subtype in anal canal
3. Anal dysplasia cytologic grade
4. Questionnaire responses
5. Adverse effects experienced during treatment, recorded in symptom log

DETAILED DESCRIPTION:
There are no further details to describe regarding this research project

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosed with perianal condyloma by primary clinician
* HIV-infected, may be on or off of antiretroviral therapy
* any CD4 count will be considered appropriate for study
* Blood WBC > 2.0x103/mm3 and absolute neutrophils count > 500
* Blood hemoglobin > 10.0 g/dL
* Blood platelet count > 50x103/mm3
* Serum total bilirubin < 6.0 mg/dL (participants taking atazanavir-based ARV regimens may have elevated total bilirubin but are generally < 6)
* Blood aspartate aminotransferase (AST) < 100 U/L (<2 ULN)
* Blood alanine aminotransferase (ALT) < 130 U/L (<2 ULN)
* Serum creatinine < 1.5 mg/dL
* ECOG performance status < 3
* If a subject is of reproductive potential he/she and her/his sexual partner MUST be willing and able to utilize effective methods of contraception (e.g., birth control pill, barrier methods with spermicide - as applicable) for the duration of the study including the study follow-up period.

Exclusion Criteria:

* Anal cancer (current or history of)
* Inability to attend study visits
* Participation in any other drug study
* History of asthma
* History of organ transplantation or requiring chronic administration of immune suppressive drugs in the last 6 months
* For women, neither pregnant nor lactating
* In the opinion of the PI, the subject may not be able to tolerate the study treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Wart characterization change is being assessed | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  Perianal wart characterization includes counting the number of identified warts, the diameter measurement of each identified wart in millimeters and the photographic imaging of each identified wart during the treatment phase and the follow-up phase of the study

SECONDARY OUTCOMES:
HPV subtype identification change is being assessed | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  HPV subtype identification specimen collection from the anal canal will be conducted during the treatment phase and the follow-up phase of the study
Anal dysplasia cytologic grade change is being assessed | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  Anal dysplasia cytologic specimen collection will take place during the treatment phase and the follow-up phase of the study
Adverse effects during the treatment phase of the study are being assessed | Days 0, 4, 11, 32, 39, 70, 100, 130, 160
  Adverse effects experienced during the treatment phase of the study are recorded by the study participants in a symptoms log

CONTACTS AND LOCATIONS:
Overall Officials: John D Malone, MD, Principal Investigator — NMCSD
Locations (1):
- NMCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No